CLINICAL TRIAL: NCT03586011
Title: Which Primary Care Patients Benefit From Physical Activity on Prescription? An Analysis of Factors Predicting Increased Physical Activity
Brief Title: Predictors of Increased Physical Activity in Patients Receiving Physical Activity on Prescription
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Stefan Lundqvist, Physiotherapist, Vastra Gotaland Region
Other Study IDs: Predictor study 206151
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2019-06

CONDITIONS: Health Behavior; Physical Activity; Metabolic Syndrome X; Primary Health Care
Keywords: Physical activity on prescription; Correlate of physical activity; Predicting factor
MeSH Terms: conditions — Health Behavior; Motor Activity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Predicting factors for increased physical activity

SUMMARY:
The aim of this study is to explore possible predicting factors associated with physical activity (PA) level change in a 6-month period of physical activity on prescription (PAP) treatment. This is done in order to highlight potential predictors important for increased PA-level and to identify which primary care patients who may benefit from the PAP-intervention.

Four hundred forty four patients are included in the study, 27-85 years, physically inactive, having at least one component of the metabolic syndrome (MetS) present and receiving PAP-treatment. Possible predicting factors of PA change at baseline and PA-level at 6-month follow-up are analyzed.

DETAILED DESCRIPTION:
Aim:

To explore possible predicting factors associated with PA-level change in a 6-month period of PAP-treatment. This is done in order to highlight potential predictors important for increased PA-level and to identify which primary care patients who may benefit from the PAP-intervention.

Methods:

Study design:

This is a longitudinal prospective observational cohort study with a 6-month follow-up of PAP-treatment. The treatment is carried out as part of a daily clinical primary care practice.

Study population:

The 444 patients included in the study, are selected from 15 primary health care centres in Gothenburg, Sweden, and are 27-85 years, physically inactive, having at least one component of the MetS present and receiving PAP-treatment. The patients have to understand the Swedish language to fill in the questionnaires.

Intervention:

The PAP-treatment is offered by authorized personnel, educated in PA-effects and PAP-intervention and consists of an individual-based dialogue with the patient, an individually tailored recommendation of PA including a written prescription, and customized, structured support during 6 months. The patients health status, previous respectively current PA level, preferences for different physical activities, motivation, self-efficacy and readiness to change PA behavior are evaluated. An agreed individually dosed PA is written down and the support during the 6-month intervention is individually structured either by revisits or by telephone contacts.

Measurements:

The following measurements are conducted at baseline and the 6-month follow-up: PA-level, self-efficacy expectations, outcome expectations, enjoyment, social support, readiness to change PA, body mass index (BMI), and health related quality of life. Age, sex, social situation, economy, education, and smoking is also measured.

Statistical analysis:

A per-protocol analysis is used. In the predictor analysis, Spearman rank correlation and a univariate regression analysis is used, respectively, to examine the association between possible predicting factors at baseline and PA level at 6-month follow-up. Significant predictors from the regression analysis are dichotomized into positive and negative values, respectively, and a Chi-square test for independence is used in analysing the predictors at baseline to increased PA level at 6-month follow-up. Statistical significance is set at p ≤0.05.

Hypothesis:

It is possible finding predicting factors among the patient´s answers according to self-reported questionnaires for the purpose of identifying responders/non-responders to increased physical activity level at 6 month follow-up of PAP-treatment.

Clinical implication:

Highlighting possible predicting factors to increased PA in an early stage of PAP-intervention, offers the opportunity to support the patient in the behavioural change process and to individualize the PAP-treatment, with the aim to increase physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive according to ACSM/AHA public health recommendation from 2007.
* Having at least one component of the metS present according to the National Cholesterol Education Program (NCEP) classification.
* Receiving PAP-treatment.
* Understanding the Swedish language.

Exclusion Criteria:

* The patient decline to participate.

Ages: 27 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The 444 patients included in the study, are selected from 15 primary health care centres in Gothenburg, Sweden and are 27-85 years, physically inactive, having at least one component of the MetS present and receiving PAP-treatment. The patients have to understand the Swedish language to fill in the questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Change in self-assessed PA-level according to the public health recommendation. | Change between baseline and 6-month follow-up. Association between PA-level at 6-month follow-up and baseline value of secondary outcome.
  Self-assessment of PA-level according to American college of sports medicine (ACSM) and American heart association (AHA) public health recommendation 2007. The patient responds to two PA questions, where 30 minutes of moderate-intensity PA per day results in 1 point and 20 minutes of more vigorous-intensity PA per day results in 1.7 point during each specific day of the week. A value of <5 points indicates an inadequate PA level.

SECONDARY OUTCOMES:
Self-efficacy expectations - Self-Efficacy for Exercise Scale (SEE) | Association between baseline value of secondary outcome and 6-month value of primary outcome.
  Questionnaire focusing on the ability to exercise for 20 minutes, three times per week in the face of barriers to exercise. The questionnaire is culturally adopted, translated into Swedish, and includes nine items (e.g. "The weather was bothering you", "You had to exercise alone", "You felt depressed"), rated on an ordinal 10 point scale ranging from 1 (Not confident) to 10 (Very confident). The item scores are summarized and divided by the number of responses indicating the strength of self-efficacy expectations. The SEE has been tested for older adults and older women post-hip fracture displaying high internal consistency, acceptable reliability measured with squared multiple correlation coefficients and sufficient to strong evidence for construct- and criterion validity.
Outcome expectations - Outcome Expectations for Exercise-2 Scale (OEE-2) | Association between baseline value of secondary outcome and 6-month value of primary outcome.
  A 13-item measure with 9 positive worded items (e.g. "Helps me feel less tired") and 4 negatively worded items (e.g. "Is something I avoid because it causes me to be short of breath") divided into two subscales: positive OEE and negative OEE. The items are rated on a 5 point Likert scale ranging from 1 (Strongly agree) to 5 (Strongly disagree). The negative OEE items are reversed scored and the numerical ratings for each response are summarized and divided by the number of items. The OEE-2 questionnaire was revised in year 2005 to include 4 items concerning negative expectations with exercise based on qualitative findings and has shown some evidence for convergent validity, internal consistency and person-, item reliability.
Enjoyment - Physical Activity Enjoyment Scale (PACES) | Association between baseline value of secondary outcome and 6-month value of primary outcome.
  Consists of 16 items whereof 9 positively worded (e.g." I think it´s fun", "It gives me energy", "It is very pleasant") and 7 negatively worded (e.g. "I feel bored", "I don´t like it", "It´s frustrating for me"). Each item is rated on a 5 point Likert scale from 1 (Does not apply at all) to 5 (Truly applies), the negatively worded items are reversed scored and the responses are added to a score ranging from 16 to 80. The PACES has been tested for 18-24 year old students and adults with functional limitations showing acceptable test-retest reliability, internal consistency and criterion validity correlated to physical function.
Social support - Social support for exercise scale (SSES) | Association between baseline value of secondary outcome and 6-month value of primary outcome.
  Including 13 items, divided in a family and friends part and measured on a 5 point Likert scale. Eleven items are positively worded (participation and involvement) and two items negatively (rewards and punishments) describing social interactions possibly linked to exercise behaviour during the previous three months. Responses were ranged from 1 (none) to 5 (very often) and "not applicable" was given a score of 1. The item scores are summarized in three subgroups: Family support - positive, Friend support - positive and Family support - negative. The Friend support - negative subgroup scores were excluded by Sallis et al. because it did not emerge in the factor analysis. The SSES has shown acceptable test-retest reliability, high internal consistency and significant criterion validity correlated with a vigorous exercise measure.
The readiness to change PA level | Association between baseline value of secondary outcome and 6-month value of primary outcome.
  Measured at baseline including three questions estimated on a 100 mm visual analogue scale (VAS): How prepared are you? How important is it for you? How confident are you to succeed (self-efficacy)? The VAS line is anchored in each ends with words describing the minimal respectively maximal extremes of the dimension being measured. The questions derives from MI and behaviour change counselling according to Rollnick et al where a higher value on the VAS indicates increased readiness to change. VAS has been used in the social and behavior sciences both as a research and clinical tool and is considered to have acceptable reliability and validity.
Body mass index - BMI | Association between baseline value of secondary outcome and 6-month value of primary outcome.
  Calculated (kg/m2) from measured body weight, with light clothing and without shoes to the nearest 0.1 kg using an electric scale (Carl Lidén AFW D300, Jönköping, Sweden) and body height, measured in an upright position without shoes to the nearest 0.5 cm using a scale fixed to the wall (PEM 136, Hultafors, Sweden).
Health related quality of life - the Swedish version of the Short Form 36 (SF-36 Standard Swedish Version 1.0) | Association between baseline value of secondary outcome and 6-month value of primary outcome.
  Includes 36 questions and generates eight health concepts: physical functioning (PF), role physical functioning (RP), bodily pain (BP), general health (GH), vitality (VT), social function (SF), role emotional functioning (RE) and mental health (MH). The health concepts are converted to 0-100 points where higher values represents a better health-related quality of life. The different health concepts of SF-36 are also grouped into a physical component summary (PCS) and mental component summary (MCS) respectively. SF-36 has shown good to excellent internal consistency reliability and is validated in a representative sample of Swedish population.
Socio demographic data. | Association between baseline value of secondary outcome and 6-month value of primary outcome.
  Age (years), sex (female-male), social situation (single-married/cohabit-other), economy (good-neither nor-bad), education (elementary grade-upper secondary school-university college) and smoking (yes-previous-no) were also measured.

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Cider, PhD, Principal Investigator — Department of Health and Rehabilitation, Unit of Physiotherapy, Institute of Neuroscience and Physiology, Sahlgrenska Academy, University of Gothenburg, , Gothenburg, Sweden
Locations (1):
- Närhälsan Göteborg centrum för fysisk aktivitet, Gothenburg, Region Västra Götaland, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Unidentifiable patient data for all primary and secondary outcome measures will be made available in a source data file (XLSX) in published article.
Time Frame: A source data file will be available in section "Supporting information" in published article.

REFERENCES:
- [Background] Das P, Horton R. Rethinking our approach to physical activity. Lancet. 2012 Jul 21;380(9838):189-90. doi: 10.1016/S0140-6736(12)61024-1. No abstract available. PMID 22818931
- [Background] Grundy SM, Brewer HB Jr, Cleeman JI, Smith SC Jr, Lenfant C; American Heart Association; National Heart, Lung, and Blood Institute. Definition of metabolic syndrome: Report of the National Heart, Lung, and Blood Institute/American Heart Association conference on scientific issues related to definition. Circulation. 2004 Jan 27;109(3):433-8. doi: 10.1161/01.CIR.0000111245.75752.C6. No abstract available. PMID 14744958
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Wen CP, Wai JP, Tsai MK, Yang YC, Cheng TY, Lee MC, Chan HT, Tsao CK, Tsai SP, Wu X. Minimum amount of physical activity for reduced mortality and extended life expectancy: a prospective cohort study. Lancet. 2011 Oct 1;378(9798):1244-53. doi: 10.1016/S0140-6736(11)60749-6. Epub 2011 Aug 16. PMID 21846575
- [Background] Hagberg LA, Lindahl B, Nyberg L, Hellenius ML. Importance of enjoyment when promoting physical exercise. Scand J Med Sci Sports. 2009 Oct;19(5):740-7. doi: 10.1111/j.1600-0838.2008.00844.x. Epub 2008 Aug 5. PMID 18694433
- [Background] Joy EL, Blair SN, McBride P, Sallis R. Physical activity counselling in sports medicine: a call to action. Br J Sports Med. 2013 Jan;47(1):49-53. doi: 10.1136/bjsports-2012-091620. Epub 2012 Nov 13. PMID 23149653
- [Background] Persson G, Brorsson A, Ekvall Hansson E, Troein M, Strandberg EL. Physical activity on prescription (PAP) from the general practitioner's perspective - a qualitative study. BMC Fam Pract. 2013 Aug 29;14:128. doi: 10.1186/1471-2296-14-128. PMID 23987804
- [Background] Sallis R, Franklin B, Joy L, Ross R, Sabgir D, Stone J. Strategies for promoting physical activity in clinical practice. Prog Cardiovasc Dis. 2015 Jan-Feb;57(4):375-86. doi: 10.1016/j.pcad.2014.10.003. Epub 2014 Oct 22. PMID 25459975
- [Background] Bauman AE, Sallis JF, Dzewaltowski DA, Owen N. Toward a better understanding of the influences on physical activity: the role of determinants, correlates, causal variables, mediators, moderators, and confounders. Am J Prev Med. 2002 Aug;23(2 Suppl):5-14. doi: 10.1016/s0749-3797(02)00469-5. PMID 12133733
- [Background] Baranowski T, Anderson C, Carmack C. Mediating variable framework in physical activity interventions. How are we doing? How might we do better? Am J Prev Med. 1998 Nov;15(4):266-97. doi: 10.1016/s0749-3797(98)00080-4. PMID 9838973
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Bauman AE, Reis RS, Sallis JF, Wells JC, Loos RJ, Martin BW; Lancet Physical Activity Series Working Group. Correlates of physical activity: why are some people physically active and others not? Lancet. 2012 Jul 21;380(9838):258-71. doi: 10.1016/S0140-6736(12)60735-1. PMID 22818938
- [Background] Stott NC, Rollnick S, Rees MR, Pill RM. Innovation in clinical method: diabetes care and negotiating skills. Fam Pract. 1995 Dec;12(4):413-8. doi: 10.1093/fampra/12.4.413. PMID 8826057
- [Background] Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000 May-Jun;49(3):154-9. doi: 10.1097/00006199-200005000-00007. PMID 10882320
- [Background] Resnick B. Reliability and validity of the Outcome Expectations for Exercise Scale-2. J Aging Phys Act. 2005 Oct;13(4):382-94. doi: 10.1123/japa.13.4.382. PMID 16301750
- [Background] Motl RW, Dishman RK, Saunders R, Dowda M, Felton G, Pate RR. Measuring enjoyment of physical activity in adolescent girls. Am J Prev Med. 2001 Aug;21(2):110-7. doi: 10.1016/s0749-3797(01)00326-9. PMID 11457630
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Allender S, Hutchinson L, Foster C. Life-change events and participation in physical activity: a systematic review. Health Promot Int. 2008 Jun;23(2):160-72. doi: 10.1093/heapro/dan012. Epub 2008 Mar 25. PMID 18364364
- [Background] Kallings LV, Sierra Johnson J, Fisher RM, Faire Ud, Stahle A, Hemmingsson E, Hellenius ML. Beneficial effects of individualized physical activity on prescription on body composition and cardiometabolic risk factors: results from a randomized controlled trial. Eur J Cardiovasc Prev Rehabil. 2009 Feb;16(1):80-4. doi: 10.1097/HJR.0b013e32831e953a. PMID 19237997
- [Background] Leijon ME, Bendtsen P, Nilsen P, Festin K, Stahle A. Does a physical activity referral scheme improve the physical activity among routine primary health care patients? Scand J Med Sci Sports. 2009 Oct;19(5):627-36. doi: 10.1111/j.1600-0838.2008.00820.x. Epub 2008 Jul 8. PMID 18627557
- [Background] Olsson SJ, Borjesson M, Ekblom-Bak E, Hemmingsson E, Hellenius ML, Kallings LV. Effects of the Swedish physical activity on prescription model on health-related quality of life in overweight older adults: a randomised controlled trial. BMC Public Health. 2015 Jul 21;15:687. doi: 10.1186/s12889-015-2036-3. PMID 26193882
- [Background] Rodjer L, H Jonsdottir I, Borjesson M. Physical activity on prescription (PAP): self-reported physical activity and quality of life in a Swedish primary care population, 2-year follow-up. Scand J Prim Health Care. 2016 Dec;34(4):443-452. doi: 10.1080/02813432.2016.1253820. Epub 2016 Nov 20. PMID 27978781
- [Background] Dwamena F, Holmes-Rovner M, Gaulden CM, Jorgenson S, Sadigh G, Sikorskii A, Lewin S, Smith RC, Coffey J, Olomu A. Interventions for providers to promote a patient-centred approach in clinical consultations. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD003267. doi: 10.1002/14651858.CD003267.pub2. PMID 23235595
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Sullivan M, Karlsson J, Ware JE Jr. The Swedish SF-36 Health Survey--I. Evaluation of data quality, scaling assumptions, reliability and construct validity across general populations in Sweden. Soc Sci Med. 1995 Nov;41(10):1349-58. doi: 10.1016/0277-9536(95)00125-q. PMID 8560302
- [Background] McCormack HM, Horne DJ, Sheather S. Clinical applications of visual analogue scales: a critical review. Psychol Med. 1988 Nov;18(4):1007-19. doi: 10.1017/s0033291700009934. PMID 3078045
- [Background] Keys A, Fidanza F, Karvonen MJ, Kimura N, Taylor HL. Indices of relative weight and obesity. J Chronic Dis. 1972 Jul 1;25(6):329-43. doi: 10.1016/0021-9681(72)90027-6. No abstract available. PMID 4650929
- [Background] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Result] Lundqvist S, Borjesson M, Larsson ME, Hagberg L, Cider A. Physical Activity on Prescription (PAP), in patients with metabolic risk factors. A 6-month follow-up study in primary health care. PLoS One. 2017 Apr 12;12(4):e0175190. doi: 10.1371/journal.pone.0175190. eCollection 2017. PMID 28403151
- [Derived] Lundqvist S, Borjesson M, Larsson MEH, Cider A, Hagberg L. Which patients benefit from physical activity on prescription (PAP)? A prospective observational analysis of factors that predict increased physical activity. BMC Public Health. 2019 May 2;19(1):482. doi: 10.1186/s12889-019-6830-1. PMID 31046720